CLINICAL TRIAL: NCT06860438
Title: Can Perfusion Index Indicate the Need of Vasopressor in ICU Patients with Sepsis and Septic Shock, Prospective Observational Study
Brief Title: Observational Study About the Use of Perfusion Index to Use Vasopressor in Sepsis
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nancy shaker shaker elhusseiny, Assistant lecturer of anesthesia, Ain Shams University
Other Study IDs: FMASU MD12/2024
Record Dates: First submitted 2025-02-17; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Perfusion Index; Vasopressor
MeSH Terms: conditions — Sepsis | interventions — Vasoconstrictor Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- vasopressor
  Interventions: Drug: Vasoconstrictor Agents
- no vasopressor

INTERVENTIONS:
Drug: Vasoconstrictor Agents — vasopressor agents will be started in patients with sepsis who will not improved using the resuscitation fluids
  Groups: vasopressor

SUMMARY:
In this thesis we will use the current state of knowledge that PI can provide a reliable information about the state of peripheral microcirculation during the state of sepsis and septic shock in ICU patients and that can interfere with the timing of starting vasopressor treatment in sepsis and septic shock

DETAILED DESCRIPTION:
Septic shock is the leading cause of death worldwide, with in-hospital and intensive care mortality rates of 11.9% to 47.2%, depending on the setting and severity of the disease .

Endothelial dysfunction is a key element in sepsis pathophysiology. It is responsible for the sepsis-induced hypotension. So the essential step in the management of sepsis is to increase systemic and regional/microcirculatory flow. Increasing arterial blood pressure (ABP) with vasopressors when patients are hypotensive is used to improve the input pressure driving organ perfusion .

Experts' recommendations currently position norepinephrine (NE) as the first-line vasopressor in septic shock. Its early administration may allow achieving the initial mean arterial pressure (MAP) target faster and reducing the risk of fluid overload. However , controversies still exist on some issues such as, whether very early use of norepinephrine (NE) could improve outcome, whether individualized target of mean arterial pressure (MAP) should be applied . Perfusion index (PI) is a reliable noninvasive indicator of peripheral perfusion derived from the photoelectric plethysmographic (PPG) signal of a pulse oximetry . The perfusion index (PI) represents the ratio of pulsatile on non-pulsatile light absorbance or reflectance of the PPG signal. PI determinants are complex and interlinked, involving and reflecting the interaction between peripheral and central hemodynamic characteristics, such as vascular tone and stroke volume. Recently, several studies have shed light on the interesting performances of this variable, especially assessing hemodynamic monitoring in anesthesia, perioperative and intensive care.

Peripheral perfusion index is an early predictor of central hypovolemia. In a prospective observational study in an emergency department, PPI was not significantly different between patients admitted to the hospital and patients discharged from the emergency department suggesting that it could not be used as a triage tool . However, Lime A with his colleagues found that PPI is significantly lower in critically ill patients with a peripheral perfusion alteration(0.7 vs 2.3, p < 0.01) Another study showed that the PPI is altered in septic shock patients, as compared to control subjects in postoperative scheduled surgery. Moreover, in the same study, the PPI was significantly lower in non-survivors. With a 0.20 cutoff value, PPI was predictive of ICU mortality with an AUC of 84% (69-96), a sensitivity of 65% and a specificity of 92%.

ELIGIBILITY:
Inclusion Criteria:

- All ICU patients with clinically suspected sepsis and septic shock ( signs include fever hypotension oliguria and confusion combined with culture results showing infection .Septic shock is a subset of sepsis involves persistent hypotension (mean arterial pressure ≥ 65 mm Hg, and a serum lactate level > 18 mg/dL [2 mmol/L)not responding to fluid resuscitation ) .

Exclusion Criteria:

* Pregnant females
* Patients on vasopressor or positive inotropic drugs
* Patients with hypothermia (defined as central temperature <35°C).
* Patient with impairment of upper extremity circulation,(such as those who underwent radial artery harvesting for coronary artery bypass grafting or had suspected occlusion of the radial artery prior to surgery,)
* Patients had undergone an operation that involved the large arteries of the aortic arch.
* Patients with atherosclerosis .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with sepsis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
PI (perfusion index ) variable will be measured at the start of resuscitation and at the start of vasopressor therapy | PI variable will be recorded at baseline( T0 )and after 5 minutes from starting of resuscitation (T5) and then 6 hours thereafter for 24 hours
  PI will be measured at the start of resuscitation after volume resuscitation and before the use of vasopressor then will be measured 6 hours after resuscitation

SECONDARY OUTCOMES:
Mean arterial Blood pressure | Baseline (T0 ) ,5 miutes after initial fluid resuscitation (T5) and 6 hours thereafter (T6) for 24 hours
  mean arterial blood pressure in mmHg
Heart rate (HR) | Baseline (T0 ) ,5 miutes after initial fluid resuscitation (T5) and 6 hours thereafter (T6) for 24 hours
  in beat per minute (bpm)
The central venous-arterial blood carbon dioxide partial pressure difference (Pv-aCO2) | Baseline (T0 ) ,5 minutes after initial fluid resuscitation (T5) and 6 hours thereafter (T6) for 24 hours
  The central venous-arterial blood carbon dioxide partial pressure difference (Pv-aCO2) will be calculated as the difference between the partial pressures of central venous carbon dioxide (PcvCO2) and arterial carbon dioxide (PaCO2).
arterial lactate concentration | Baseline (T0 ) ,5 minutes after initial fluid resuscitation (T5) and 6 hours thereafter (T6) for 24 hours
ScvO2 (central venous oxygen saturation ) | Baseline (T0 ) ,5 minutes after initial fluid resuscitation (T5) and 6 hours thereafter (T6) for 24 hours
  ScvO2 will be calculated from a sample taken from the central venous catheter.
APACHE Score | first 24 hours
  APACHE score stands for acute physiology and chronic health evaluation.APACHE scores use clinical, physiological and laboratory data observed at admission and during the first 24 hours after ICU admission. This is in order to estimate a given patient's severity of illness by providing a severity score and a probability of hospital death .It consists of twelve acute physiologic variables, age, and chronic health status. The APACHE II score is determined by totalling points from these three sections, resulting in a total score between 0 and 71 points (0 is low risk and 71 is the high risk )
SOFA score | 48 hours
  SOFA score stands for Sequential Organ Failure Assessment .it is a composite score based on the degree of dysfunction in six organ systems-respiratory, coagulation, hepatic, cardiovascular, central nervous system, and renal . Each organ dysfunction scores from 0 to 4, with increasing scores reflecting more abnormal physiology and biochemistry or an increasing degree of intervention Score ranges from 0 (best) to 24 (worst) points
Mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Nancy shaker ass,lecurer, Principal Investigator — faculty of medicine, Ain Shams University
Locations (1):
- faculty of medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No